CLINICAL TRIAL: NCT00336284
Title: TRUST: Lumos-T Safely RedUceS RouTine Office Device Follow-up
Acronym: TRUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Justin Michalski, M.S. / Clinical Studies Engineer, BIOTRONIK, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20052069
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Patient Indicated for an ICD
Keywords: Telemonitoring; ICD; Reduction of office follow-ups
MeSH Terms: interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Monitoring (Active Comparator): Home Monitoring programmed on.
  Interventions: Other: Home Monitoring
- In-Office Conventional Follow-up (Other): Home Monitoring programmed off.
  Interventions: Other: In-Office Conventional Follow-up

INTERVENTIONS:
Other: Home Monitoring — Home Monitoring programmed on. In-office and Home Monitoring evaluation at 3 and 15 months post ICD implant. Home Monitoring evaluation only at 6, 9, and 12 months post ICD implant.
  Arms: Home Monitoring
Other: In-Office Conventional Follow-up — Home Monitoring programmed off. In-office evaluations at 3, 6, 9, 12, and 15 months post ICD implant.
  Arms: In-Office Conventional Follow-up

SUMMARY:
This study is a multi-center, prospective and randomized trial. The primary objective of this study is to demonstrate that the use of the BIOTRONIK Home Monitoring system (HM) can safely reduce the number of regularly scheduled office follow-up visits, compared to the conventional method of implantable cardioverter defibrillator (ICD) follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Implanted within the last 45 days or being considered for implant with a BIOTRONIK ICD with Home Monitoring (HM)/Intracardiac Electrogram (IEGM)-Online technology, or legally marketed future generation device with HM/IEGM Online.
* Able to utilize the HM system throughout the study
* Ability to give informed consent
* Geographically stable and able to return for regular follow-ups for fifteen (15) months
* At least 18 years old

Exclusion Criteria:

* Patients who do not fulfill all inclusion criteria
* Pacemaker dependent
* Currently enrolled in any other cardiac clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Actual)
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Varma, MD, FRCP, Principal Investigator — The Cleveland Clinic
Locations (110):
- United States (108):
  - Site 55, Birmingham, Alabama
  - Site 68, Mesa, Arizona
  - Site 99, Phoenix, Arizona
  - Site 118, Bakersfield, California
  - Site 91, Bakersfield, California
  - Site 95, Burbank, California
  - Site 72, Fairfield, California
  - Site 43, Fremont, California
  - Site 90, Fresno, California
  - Site 73, Fresno, California
  - Site 75, Fresno, California
  - Site 67, Glendale, California
  - Site 82, Jackson, California
  - Site 78, Mission Viejo, California
  - Site 15, Sherman Oaks, California
  - Site 89, Simi Valley, California
  - Site 88, Whittier, California
  - Site 37, Boulder, Colorado
  - Site 38, Boulder, Colorado
  - Site 98, Denver, Colorado
  - Site 122, Newark, Delaware
  - Site 100, Brooksville, Florida
  - Site 111, Jacksonville, Florida
  - Site 40, Lakeland, Florida
  - Site 36, Lauderdale Lakes, Florida
  - Site 34, Miami, Florida
  - Site 42, Oakland Park, Florida
  - Site 13, Port Charlotte, Florida
  - Site 41, Tamarac, Florida
  - Site 60, Vero Beach, Florida
  - Site 6, Canton, Georgia
  - Site 106, Douglas, Georgia
  - Site 61, Lawrenceville, Georgia
  - Site 10, Marietta, Georgia
  - Site 66, Marietta, Georgia
  - Site 21, Chicago, Illinois
  - Site 124, Chicago, Illinois
  - Site 39, Oak Lawn, Illinois
  - Site 3, Louisville, Kentucky
  - Site 11, Owensboro, Kentucky
  - Site 51, Covington, Louisiana
  - Site 79, Hammond, Louisiana
  - Site 85, Lacombe, Louisiana
  - Site 102, Lafayette, Louisiana
  - Site 2, Lake Charles, Louisiana
  - Site 53, New Orleans, Louisiana
  - Site 17, Annapolis, Maryland
  - Site 25, Lanham, Maryland
  - Site 17, Riverdale, Maryland
  - Site 18, Rockville, Maryland
  - Site 29, Boston, Massachusetts
  - Site 94, Ann Arbor, Michigan
  - Site 103, Bloomfield Hills, Michigan
  - Site 4, Lansing, Michigan
  - Site 12, Lapeer, Michigan
  - Site 22, Saginaw, Michigan
  - Site 14, Corinth, Mississippi
  - Site 52, Gulfport, Mississippi
  - Site 49, Bridgeton, Missouri
  - Site 105, Festus, Missouri
  - Site 121, Festus, Missouri
  - Site 45, Moberly, Missouri
  - Site 56, Osage Beach, Missouri
  - Site 108, St Louis, Missouri
  - Site 114, St Louis, Missouri
  - Site 48, St Louis, Missouri
  - Site 113, St Louis, Missouri
  - Site 74, St Louis, Missouri
  - Site 47, University City, Missouri
  - Site 117, Brick, New Jersey
  - Site 120, East Brunswick, New Jersey
  - Site 107, East Orange, New Jersey
  - Site 119, Elizabeth, New Jersey
  - Site 116, Oakhurst, New Jersey
  - Site 71, Wayne, New Jersey
  - Site 97, Las Cruces, New Mexico
  - Site 112, Batavia, New York
  - Site 19, Brooklyn, New York
  - Site 27, Brooklyn, New York
  - Site 26, Brooklyn, New York
  - Site 77, Brooklyn, New York
  - Site 9, Johnson City, New York
  - Site 35, New York, New York
  - Site 76, New York, New York
  - Site 115, Pinehurst, North Carolina
  - Site 57, Cleveland, Ohio
  - Site 16, Columbus, Ohio
  - Site 50, Columbus, Ohio
  - Site 84, Fairview Park, Ohio
  - Site 93, Massillon, Ohio
  - Site 30, Middletown, Ohio
  - Site 87, Middletown, Ohio
  - Site 96, Tulsa, Oklahoma
  - Site 63, Chinchilla, Pennsylvania
  - Site 62, Clarks Summit, Pennsylvania
  - Site 32, Upland, Pennsylvania
  - Site 23, Columbia, South Carolina
  - Site 20, Florence, South Carolina
  - Site 109, Lancaster, South Carolina
  - Site 5, Rock Hill, South Carolina
  - Site 59, Knoxville, Tennessee
  - Site 8, Knoxville, Tennessee
  - Site 110, Tullahoma, Tennessee
  - Site 1, Amarillo, Texas
  - Site 81, Brownsville, Texas
  - Site 33, Odessa, Texas
  - Site 80, San Antonio, Texas
  - Site 7, Yakima, Washington
- Canada (2):
  - Site 104, Toronto, Ontario
  - Site 92, Fleurimont, Quebec

REFERENCES:
- [Result] Varma N, Epstein AE, Irimpen A, Schweikert R, Love C; TRUST Investigators. Efficacy and safety of automatic remote monitoring for implantable cardioverter-defibrillator follow-up: the Lumos-T Safely Reduces Routine Office Device Follow-up (TRUST) trial. Circulation. 2010 Jul 27;122(4):325-32. doi: 10.1161/CIRCULATIONAHA.110.937409. Epub 2010 Jul 12. PMID 20625110
- [Derived] Chew DS, Piccini JP, Au F, Frazier-Mills CG, Michalski J, Varma N; TRUST Investigators. Alert-driven vs scheduled remote monitoring of implantable cardiac defibrillators: A cost-consequence analysis from the TRUST trial. Heart Rhythm. 2023 Mar;20(3):440-447. doi: 10.1016/j.hrthm.2022.12.003. Epub 2022 Dec 8. PMID 36503177
- [Derived] Varma N, Love CJ, Michalski J, Epstein AE; TRUST Investigators. Alert-Based ICD Follow-Up: A Model of Digitally Driven Remote Patient Monitoring. JACC Clin Electrophysiol. 2021 Aug;7(8):976-987. doi: 10.1016/j.jacep.2021.01.008. Epub 2021 Feb 24. PMID 33640345
- [Derived] Varma N, Love CJ, Schweikert R, Moll P, Michalski J, Epstein AE; TRUST Investigators. Automatic remote monitoring utilizing daily transmissions: transmission reliability and implantable cardioverter defibrillator battery longevity in the TRUST trial. Europace. 2018 Apr 1;20(4):622-628. doi: 10.1093/europace/eux059. PMID 29016878
- [Derived] Varma N, Epstein AE, Schweikert R, Michalski J, Love CJ; TRUST Investigators. Role of Automatic Wireless Remote Monitoring Immediately Following ICD Implant: The Lumos-T Reduces Routine Office Device Follow-Up Study (TRUST) Trial. J Cardiovasc Electrophysiol. 2016 Mar;27(3):321-6. doi: 10.1111/jce.12895. Epub 2016 Jan 27. PMID 26661687
- [Derived] Varma N, Michalski J, Stambler B, Pavri BB; TRUST Investigators. Superiority of automatic remote monitoring compared with in-person evaluation for scheduled ICD follow-up in the TRUST trial - testing execution of the recommendations. Eur Heart J. 2014 May 21;35(20):1345-52. doi: 10.1093/eurheartj/ehu066. Epub 2014 Mar 3. PMID 24595864
- [Derived] Varma N, Pavri BB, Stambler B, Michalski J; TRUST Investigators. Same-day discovery of implantable cardioverter defibrillator dysfunction in the TRUST remote monitoring trial: influence of contrasting messaging systems. Europace. 2013 May;15(5):697-703. doi: 10.1093/europace/eus410. Epub 2012 Dec 19. PMID 23258817
- [Derived] Varma N, Michalski J, Epstein AE, Schweikert R. Automatic remote monitoring of implantable cardioverter-defibrillator lead and generator performance: the Lumos-T Safely RedUceS RouTine Office Device Follow-Up (TRUST) trial. Circ Arrhythm Electrophysiol. 2010 Oct;3(5):428-36. doi: 10.1161/CIRCEP.110.951962. Epub 2010 Aug 17. PMID 20716717

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional: Home Monitoring programmed OFF
Period: Overall Study
Arm/Group | Home Monitoring | Conventional
Started | 977 | 473
Completed | 741 | 322
Not Completed | 236 | 151
Not completed — Death | 52 | 26
Not completed — Lost to Follow-up | 82 | 61
Not completed — Withdrawal by Physician or Subject | 102 | 64

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Monitoring | Conventional | Total
Number analyzed (Participants) | 908 | 431 | 1339
Age Continuous [Mean (Standard Deviation); unit: years] — Only participants who completed at least one follow-up visit are included in the analyses. Home Monitoring Arm, N=908; Conventional Arm, N=431.
  years | 63 (13) | 64 (12) | 64 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Only participants who completed at least one follow-up visit are included in the analyses. Home Monitoring Arm, N=908; Conventional Arm, N=431.
  Participants
    Female | 254 | 116 | 370
    Male | 654 | 315 | 969
Region of Enrollment [Number; unit: participants] — Only participants who completed at least one follow-up visit are included in the analyses. Home Monitoring Arm, N=908; Conventional Arm, N=431.
  participants
    United States | 896 | 425 | 1321
    Canada | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Home Monitoring Effectiveness
Description: Average number of office-based implantable cardioverter defibrillator (ICD) follow-up visits in the Home Monitoring arm vs the Conventional (calendar-based) follow-up arm.
Time Frame: 12 months
Population: Only participants who completed at least one follow-up visit are included in the analyses.
Measure: Mean (Full Range); unit: In-office ICD follow-up per patient year
Arm/Group | Home Monitoring | Conventional
Number analyzed (Participants) | 908 | 431
In-office ICD follow-up per patient year | 2.1 [0 to 45.6] | 3.8 [0 to 19.2]
Statistical Analysis 1: Comparison: Home Monitoring vs Conventional; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Percent of Participants Experiencing Death, Incidence of Stroke, or Event Requiring Surgical Intervention.
Description: Percentage of participants experiencing death, incidence of stroke, or event(s) requiring surgical intervention. Outcome measure time frame is 12 months.
Time Frame: 12 months
Population: Safety Event Rate includes events occuring within 12 months of enrollment for participants with at least 1 follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | Home Monitoring | Conventional
Number analyzed (Participants) | 908 | 431
Percentage of participants | 10.4 | 10.4
Statistical Analysis 1: Comparison: Home Monitoring vs Conventional; Test type: Non-Inferiority or Equivalence — Sample size of the study is based on the safety endpoint and based on a Blackwelder type test of non inferiority with the standard design criteria: Type I error (one-sided), statistical power of 80%, and 2:1 randomization. The evaluation of the primary safety endpoint was based on an exact binomial non-inferiority test comparing the proportions of patient deaths, strokes or surgical interventions; p = 0.005, Exact binomial test for non-inferiority; 1-sided

3. Secondary Outcome: Early Detection of Cardiac Events
Description: Detection time relative to onset of cardiac events (atrial fibrillation, ventricular tachycardia, ventricular fibrillation).
Time Frame: 12 months
Population: Only participants with at least one follow-up are included in the analyses.
Measure: Mean (Full Range); unit: Days
Arm/Group | Home Monitoring | Conventional
Number analyzed (Participants) | 908 | 431
Days | 13.98 [0 to 256] | 45.34 [0 to 287]
Statistical Analysis 1: Comparison: Home Monitoring vs Conventional; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

4. Secondary Outcome: Patient Initiated Follow-up
Description: Percentage of total patient initiated inqueries that result in ER or office follow-up visits.
Time Frame: 12 months
Population: Only participants with at least one follow-up are included in the analyses
Measure: Number; unit: percent of patient initiated follow-ups
Arm/Group | Home Monitoring | Conventional
Number analyzed (Participants) | 908 | 431
percent of patient initiated follow-ups | 92.7 | 100

ADVERSE EVENTS:
Time Frame: 15 Months
Description: Strokes or complications that lead to a surgical intervention were required to be reported. Complications that led to a surgical intervention include but are not limited to a lead revision, cardiac interventional procedure, or device replacement. Other AEs were reported at the discretion of the investigator and may include non-cardiac events.
Arm/Group | Home Monitoring | Conventional
Serious Adverse Events (participants affected / at risk) | 124/977 | 74/473
Other Adverse Events (participants affected / at risk) | 0/977 | 0/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Monitoring (N=977) | Conventional (N=473)
Ablation procedure (Surgical and medical procedures) | 5 (5) | 4 (4)
Aborted upgrade procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac related hospitalizations (Cardiac disorders) | 45 (64) | 31 (35)
Catheterization/PCI procedure (Surgical and medical procedures) | 15 (16) | 3 (4)
Coronary artery bypass graft procedure (Surgical and medical procedures) | 3 (3) | 0 (0)
Death (General disorders) | 52 (52) | 26 (26)
Device change-out (Surgical and medical procedures) | 8 (8) | 3 (3)
Device revision (Surgical and medical procedures) | 17 (18) | 7 (7)
Heart transplant (Surgical and medical procedures) | 1 (1) | 0 (0)
IVC filter implanted (Surgical and medical procedures) | 1 (1) | 0 (0)
LV assist device implanted (Surgical and medical procedures) | 1 (1) | 0 (0)
Lead revision/explant/replacement (Surgical and medical procedures) | 16 (16) | 5 (5)
Non-cardiac related hospitalizations (General disorders) | 16 (20) | 3 (4)
Non-cardiac surgical interventions (Surgical and medical procedures) | 7 (8) | 3 (4)
Permacath for dialysis and endoscopy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tighten loose set screw (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide copies of any abstracts, papers or manuscripts to the Sponsor for review within a reasonable period prior to submittal for publication. BIOTRONIK limits its review to a determination of whether Confidential Information (CI) is disclosed and may not attempt to censor or in any way interfere with the investigator's presentation or conclusions beyond the extent necessary to protect CI or to allow to protect its rights in patentable or copyrightable material.